CLINICAL TRIAL: NCT00090181
Title: A Double-Blind, Parallel-group, 4-Week Trial to Assess the Efficacy and Safety of Etoricoxib 60 mg and Diclofenac 150 mg in Patients With Chronic Low Back Pain
Brief Title: Study of MK0663 in Patients With Chronic Low Back Pain (0663-806)(COMPLETED)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0663-806; 2004_003
Record Dates: First submitted 2004-08-25; First posted 2004-08-27 (Estimated); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Chronic Low Back Pain
Keywords: Arcoxia
MeSH Terms: interventions — Etoricoxib; Duration of Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0663, etoricoxib / Duration of Treatment: 4 weeks
Drug: Comparator: diclofenac / Duration of Treatment: 4 weeks

SUMMARY:
The purpose of this study is to evaluate the efficacy of MK0663 for the treatment of chronic low back pain and to investigate the overall safety and tolerability over four weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients 18 years of age or older, who have Chronic Low Back Pain after the discontinuation of their previous medication for their condition.
* Patients should have at least 3 months of Low Back Pain.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2004-06; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Lower back pain intensity
Safety and tolerability

SECONDARY OUTCOMES:
Disability questionnaire
Patient global assessment of response to therapy

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Zerbini C, Ozturk ZE, Grifka J, Maini M, Nilganuwong S, Morales R, Hupli M, Shivaprakash M, Giezek H; Etoricoxib CLBP Study Group. Efficacy of etoricoxib 60 mg/day and diclofenac 150 mg/day in reduction of pain and disability in patients with chronic low back pain: results of a 4-week, multinational, randomized, double-blind study. Curr Med Res Opin. 2005 Dec;21(12):2037-49. doi: 10.1185/030079905X75069. PMID 16368055